CLINICAL TRIAL: NCT00505375
Title: Effects of CTLA-4 Ig (Abatacept) On The Progression of Type 1 Diabetes In New Onset Subjects
Brief Title: Intravenous CTLA4-lg Treatment in Recent Onset Type 1 Diabetes Mellitus
Acronym: TN09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Juvenile Diabetes Research Foundation (Other); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN09 CTLA; U01DK061055 (NIH); UC4DK097835 (NIH)
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: CTLA4-Ig; Abatacept; Beta-cell function; T-cells; DPT-1; treatment; treatment of type 1 diabetes; new onset type 1 diabetes; juvenile diabetes; T1D; diabetes mellitus; Type 1 diabetes TrialNet; TrialNet
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Intravenous infusions of CTLA-4 Ig
  Interventions: Drug: CTLA-4 Ig
- 2 (Placebo Comparator): Intravenous infusions of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CTLA-4 Ig — Intravenous infusion of 10 mg/kg of CTLA-4 Ig every other week for the first two doses and then every 28 days for a total of 27 doses
  Other Names: Abatacept
  Arms: 1
Other: Placebo — Intravenous infusions of placebo every other week for the first two doses and then every 28 days for a total of 27 doses
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether treatment with CTLA4-Ig (Abatacept) in individuals with new onset T1DM will improve insulin secretion (C-peptide production) compared to placebo.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is a T-cell mediated autoimmune disease in which insulin-producing beta cells are completely or near completely destroyed resulting in life-long dependence on exogenous insulin.

CTLA4-Ig (Abatacept) inhibits a crucial stimulatory pathway in the activation of T cells. By this mechanism, the drug is thought to arrest or slow the T cell mediated autoimmune destruction of beta-cells and preserve their function. At the time of clinical onset of T1DM, a significant amount of insulin producing beta cells are destroyed, but as many as 10-20% are still capable of insulin production. By using CTLA4-Ig close to the onset of T1DM, we hope to arrest or slow down the autoimmune destruction of these beta-cells and extend the endogenous insulin production. CTLA4-Ig regulates T cell function but does not deplete T cells. Therefore, its safety profile appears to be better than other immunosuppressive agents.

Eligible participants will be randomized to the experimental or control groups. The experimental group will receive intravenous infusions of CTLA-4 Ig. The first infusion will occur at the time of randomization, followed by another infusion 2 and 4 weeks later. Subsequent infusions will be given monthly for two years during the treatment phase of the study. There is a total of 27 infusions during the treatment phase of the study.

Participants in the control group will receive intravenous infusions of placebo according to the same schedule outlined above.

Both groups will receive standard intensive diabetes treatment with insulin and dietary management.

All participants randomized into the study will be seen at study site monthly for 24 months and then every 6 months for up to an additional 2 years. Participants will undergo assessments of their insulin production, immunologic status, overall health and well being and diabetes care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-45
2. Within 3 months (100 days) of diagnosis of T1DM based on ADA criteria
3. At least one diabetes-related autoantibody
4. Stimulated C-peptide level >0.2 pmol/ml by MMTT conducted 21 days after diagnosis of T1DM and within 37 days of randomization
5. At least three months from last live immunization received and willing to forgo live vaccinations for three months following last dose of study treatment

Exclusion Criteria:

1. Immunodeficiency, chronic lymphopenia, active infection, positive PPD result or a history of malignancy
2. Serologic evidence of current or past HIV, Hepatitis B or C
3. Pregnancy, lactation, or intention of pregnancy while on study
4. Current use of immunosuppressive agents, or medications known to influence glucose tolerance or glycemic control
5. Current participation in another T1DM treatment study

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tihamer Orban, MD, Principal Investigator — Joslin Diabetes Center; Jay Skyler, MD, Study Chair — University of Miami
Locations (13):
- United States (12):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - The Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, Naomi Berrie Diabetes Center, New York, New York
  - University of Pittsburgh, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Southwestern Medical School, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/tn09-ctla4-ig/?query=TN09
URL: https://repository.niddk.nih.gov/studies/tn09-ctla4-ig/?query=TN09

REFERENCES:
- [Background] Bach JF. Insulin-dependent diabetes mellitus as an autoimmune disease. Endocr Rev. 1994 Aug;15(4):516-42. doi: 10.1210/edrv-15-4-516. PMID 7988484
- [Background] Bretscher PA. A two-step, two-signal model for the primary activation of precursor helper T cells. Proc Natl Acad Sci U S A. 1999 Jan 5;96(1):185-90. doi: 10.1073/pnas.96.1.185. PMID 9874793
- [Background] Alegre ML, Frauwirth KA, Thompson CB. T-cell regulation by CD28 and CTLA-4. Nat Rev Immunol. 2001 Dec;1(3):220-8. doi: 10.1038/35105024. PMID 11905831
- [Background] Lenschow DJ, Zeng Y, Thistlethwaite JR, Montag A, Brady W, Gibson MG, Linsley PS, Bluestone JA. Long-term survival of xenogeneic pancreatic islet grafts induced by CTLA4lg. Science. 1992 Aug 7;257(5071):789-92. doi: 10.1126/science.1323143.
- [Background] Abrams JR, Lebwohl MG, Guzzo CA, Jegasothy BV, Goldfarb MT, Goffe BS, Menter A, Lowe NJ, Krueger G, Brown MJ, Weiner RS, Birkhofer MJ, Warner GL, Berry KK, Linsley PS, Krueger JG, Ochs HD, Kelley SL, Kang S. CTLA4Ig-mediated blockade of T-cell costimulation in patients with psoriasis vulgaris. J Clin Invest. 1999 May;103(9):1243-52. doi: 10.1172/JCI5857. PMID 10225967
- [Background] Abrams JR, Kelley SL, Hayes E, Kikuchi T, Brown MJ, Kang S, Lebwohl MG, Guzzo CA, Jegasothy BV, Linsley PS, Krueger JG. Blockade of T lymphocyte costimulation with cytotoxic T lymphocyte-associated antigen 4-immunoglobulin (CTLA4Ig) reverses the cellular pathology of psoriatic plaques, including the activation of keratinocytes, dendritic cells, and endothelial cells. J Exp Med. 2000 Sep 4;192(5):681-94. doi: 10.1084/jem.192.5.681. PMID 10974034
- [Background] Moreland LW, Alten R, Van den Bosch F, Appelboom T, Leon M, Emery P, Cohen S, Luggen M, Shergy W, Nuamah I, Becker JC. Costimulatory blockade in patients with rheumatoid arthritis: a pilot, dose-finding, double-blind, placebo-controlled clinical trial evaluating CTLA-4Ig and LEA29Y eighty-five days after the first infusion. Arthritis Rheum. 2002 Jun;46(6):1470-9. doi: 10.1002/art.10294. PMID 12115176
- [Result] Orban T, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Greenbaum CJ, Marks JB, Monzavi R, Moran A, Raskin P, Rodriguez H, Russell WE, Schatz D, Wherrett D, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet Abatacept Study Group. Co-stimulation modulation with abatacept in patients with recent-onset type 1 diabetes: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jul 30;378(9789):412-9. doi: 10.1016/S0140-6736(11)60886-6. Epub 2011 Jun 28. PMID 21719096
- [Derived] Orban T, Beam CA, Xu P, Moore K, Jiang Q, Deng J, Muller S, Gottlieb P, Spain L, Peakman M; Type 1 Diabetes TrialNet Abatacept Study Group. Reduction in CD4 central memory T-cell subset in costimulation modulator abatacept-treated patients with recent-onset type 1 diabetes is associated with slower C-peptide decline. Diabetes. 2014 Oct;63(10):3449-57. doi: 10.2337/db14-0047. Epub 2014 May 16. PMID 24834977
- See also: Related Info — http://www.diabetestrialnet.org
- See also: Related Info — http://www.jdrf.org

RESULTS

PARTICIPANT FLOW:
Groups:
- CTLA-4 Ig: Intravenous infusions of CTLA-4 Ig
  CTLA-4 Ig: Intravenous infusion of 10 mg/kg of CTLA-4 Ig every other week for the first two doses and then every 28 days for a total of 27 doses
- Placebo: Intravenous infusions of placebo
  Placebo: Intravenous infusions of placebo every other week for the first two doses and then every 28 days for a total of 27 doses
Period: Overall Study
Arm/Group | CTLA-4 Ig | Placebo
Started | 77 | 35
Completed | 73 | 30
Not Completed | 4 | 5
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Travel issues | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTLA-4 Ig | Placebo | Total
Number analyzed (Participants) | 77 | 35 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (6.9) | 13.7 (5.3) | 13.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 10 | 46
  Male | 41 | 25 | 66

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Stimulated C-peptide Curve Over the First 2 Hours of a 4 Hour Mixed Meal Tolerance Test at the 2 Year Visit
Description: The primary outcome is the area under the stimulated C-peptide curve (AUC) based on data collected at time 0 to 2 hours of a 4-hour mixed meal glucose tolerance test (MMTT) conducted at the primary endpoint visit. The timed measurements are done at: 0, 15, 30 60, 90, and 120 minutes.
Time Frame: 2 years of follow up
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Groups:
- CTLA-4 Ig: Intravenous infusions 10 mg/kg of CTLA-4 Ig every other week for the first two doses and then every 28 days for a total of 27 doses
Arm/Group | CTLA-4 Ig | Placebo
Number analyzed (Participants) | 73 | 30
nmol/L | 0.375 [0.290 to 0.465] | 0.266 [0.171 to 0.368]
Statistical Analysis 1: Comparison: CTLA-4 Ig vs Placebo; The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis; Test type: Superiority or Other; p = 0.0014, ANCOVA

ADVERSE EVENTS:
Arm/Group | CTLA-4 Ig | Placebo
Serious Adverse Events (participants affected / at risk) | 11/77 | 7/35
Other Adverse Events (participants affected / at risk) | 60/77 | 26/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTLA-4 Ig (N=77) | Placebo (N=35)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Death not associated with CTCAE term (General disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Endocrine - Other (Endocrine disorders) | 1 (1) | 0 (0)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (5) | 1 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Mood alteration- Agitation (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Pain- Head/headache (General disorders) | 0 (0) | 1 (1)
Secondary Malignancy - possibly related to cancer treatment (General disorders) | 1 (1) | 0 (0)
Intra-operative Injury - Other (Surgical and medical procedures) | 1 (1) | 0 (0)
Syndromes - Other (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTLA-4 Ig (N=77) | Placebo (N=35)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 9 (14) | 5 (12)
Constitutional Symptoms - Other (General disorders) | 5 (6) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 8 (9) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 12 (14) | 1 (2)
Endocrine - Other (Endocrine disorders) | 5 (5) | 1 (1)
Dental: teeth (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 12 (16) | 4 (4)
Infection - Other (Infections and infestations) | 28 (58) | 13 (23)
Infection with unknown ANC- Pharynx (Infections and infestations) | 1 (1) | 3 (3)
Fracture (Musculoskeletal and connective tissue disorders) | 9 (12) | 5 (5)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 2 (2)
Other AE (General disorders) | 4 (4) | 1 (1)
Pain- Head/headache (General disorders) | 1 (1) | 2 (2)
Pain - Other (General disorders) | 2 (3) | 3 (4)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 2 (2)
Flu-like syndrome (General disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No